CLINICAL TRIAL: NCT02093728
Title: A Phase I, Open-label, Single-center Study to Assess the Effect of the CYP3A4 Inhibitor Itraconazole and the CYP2C19 Inhibitor Fluconazole on the Pharmacokinetics of a 25 mg Single Oral Dose of Selumetinib (AZD6244; ARRY-142866) ( Hyd-Sulfate) in Healthy Volunteers Aged 18 to 45 Years
Brief Title: To Assess the Effect of Itraconazole and Fluconazole on the Pharmacokinetics of Selumetinib in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: D1532C00083
Record Dates: First submitted 2014-03-20; First posted 2014-03-21 (Estimated); Last update posted 2015-06-30 (Estimated); Status verified 2015-06

CONDITIONS: Solid Tumours
Keywords: Phase I, healthy, pharmacokinetics
MeSH Terms: interventions — AZD 6244; Itraconazole; Fluconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- selumetinib; itraconazole; selumetinib + itraconazole (Experimental): Volunteers will receive selumetinib 25mg alone; itraconazole 200mg pre-dosing; selumetinib 25mg and itraconazole 200mg; all adminstered by mouth as a capsule
  Interventions: Drug: selumetinib; Drug: itraconazole
- selumetinib; fluconazole; selumetinib + fluconazole (Experimental): Volunteers will receive selumetinib 25mg alone administered by mouth as a capsule; fluconazole 400mg and fluconazole 200mg pre-dosing, administered by mouth as a tablet; selumetinib 25mg and fluconazole 200mg.
  Interventions: Drug: selumetinib; Drug: fluconazole

INTERVENTIONS:
Drug: selumetinib — Volunteers will recieve single oral dose of 25mg selumetinib in sequence 1, treatment A
  Other Names: (AZD6244; ARRY-142866) ( Hyd-Sulfate)
  Arms: selumetinib; itraconazole; selumetinib + itraconazole
Drug: itraconazole — Volunteers will receive oral doses of itraconazole 200 mg twice daily on Day 1 to Day 7 in sequence 1 treatment B:
  Arms: selumetinib; itraconazole; selumetinib + itraconazole
Drug: itraconazole — Volunteers will recieve a single morning dose of 200mg itraconazole on Day 8 and twice daily doses of 200mg itraconazole on Day 8 to Day 11; sequence 1 treatment C.
  Arms: selumetinib; itraconazole; selumetinib + itraconazole
Drug: selumetinib — Volunteers willl recieve a single oral dose of 25 mg selumetinib (4 hours fasted state) on Day 8; sequence 1 treatment C.
  Other Names: (AZD6244; ARRY-142866) ( Hyd-Sulfate)
  Arms: selumetinib; itraconazole; selumetinib + itraconazole
Drug: selumetinib — Volunteers will recieve single oral dose of 25mg selumetinib in sequence 2, treatment A.
  Other Names: (AZD6244; ARRY-142866) ( Hyd-Sulfate)
  Arms: selumetinib; fluconazole; selumetinib + fluconazole
Drug: fluconazole — Volunteers will recieve a single dose of 400 mg fluconazole on Day 1 and daily doses of 200 mg fluconazole on Day 2 to Day 7; sequence 2 treatment D.
  Arms: selumetinib; fluconazole; selumetinib + fluconazole
Drug: fluconazole — Volunteers will receive a morning dose of 200mg fluconazole on Day 8 and daily doses of 200mg fluconazole on Day 8 to Day 11; sequence 2 treatment E
  Arms: selumetinib; fluconazole; selumetinib + fluconazole
Drug: selumetinib — Volunteers will receive a single dose of 25mg selumetinib (4 hours fasted state) on Day 8; sequence 2 treatment E
  Arms: selumetinib; fluconazole; selumetinib + fluconazole

SUMMARY:
Study to assess the effect of Itraconazole and Fluconazole on the pharmacokinetics of Selumetinib (AZD6244; ARRY-142866) ( Hyd-Sulfate) in Healthy Male Volunteers

DETAILED DESCRIPTION:
A Open-label, Single-center Study to Assess the Effect of the CYP3A4 Inhibitor Itraconazole and the CYP2C19 Inhibitor Fluconazole on the Pharmacokinetics of a 25 mg Single Oral Dose of Selumetinib (AZD6244; ARRY-142866) ( Hyd-Sulfate) in Healthy Volunteers

ELIGIBILITY:
Inclusion Criteria: 1. Have a body mass index (BMI) between 18 and 30 kg/m2 (inclusive) and weigh at least 50 kg and no more than 100 kg. 2. Female subjects of non-childbearing potential. 3. Have a calculated creatinine clearance (CrCL) >50 mL/min using the Cockcroft-Gault formula.

Exclusion Criteria: 1. Subjects of Japanese or non-Japanese Asian ethnicity. 2. Any one parent or grandparent (maternal or paternal) is Japanese or non-Japanese. Asian (ie, China, Taiwan, Korea, Philippines, Thailand, Vietnam and Malaysia). Asian Indians are acceptable. 3. Current or past history of central serous retinopathy or retinal vein thrombosis,intra-ocular pressure >21 mmHg or uncontrolled glaucoma. 4. Any clinically relevant abnormal findings in physical examination, hematology, clinical chemistry, urinalysis, vital signs or ECG at baseline in the opinion of the investigator.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2014-04; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics of selumetinib and N-desmethyl selumetinib by assessment of area under the plasma concentration-time curve from time zero extrapolated to infinity (AUC) | Blood samples are collected pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 12, 24, 36, 48, 72 and 96 hours post dose
  Samples taken during each of the 6 treatments

SECONDARY OUTCOMES:
Pharmacokinetics of selumetinib and N-desmethyl selumetinib by assesement of area under the plasma concentration-time from time zero to the time of the last quantifiable concentration (AUC(0-t) | Blood samples are collected pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 12, 24, 36, 48, 72 and 96 hours post dose
  Samples taken during each of the 6 treatments
Pharmacokinetics of selumetinib and N-desmethyl selumetinib by assesement of area under the plasma concentration-time curve from time zero to 12 hours post-dose AUC(0-12) | Blood samples are collected pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 12, 24, 36, 48, 72 and 96 hours post dose
  Samples taken during each of the 6 treatments
Pharmacokinetics of selumetinib and N-desmethyl selumetinib by assesement of maximum plasma concentration (Cmax) | Blood samples are collected pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 12, 24, 36, 48, 72 and 96 hours post dose
  Samples taken during each of the 6 treatments
Pharmacokinetics of selumetinib and N-desmethyl selumetinib by assesement of time to Cmax (tmax) | Blood samples are collected pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 12, 24, 36, 48, 72 and 96 hours post dose
  Samples taken during each of the 6 treatments
Pharmacokinetics of selumetinib by assesement of apparent oral plasma clearance (CL/F) | Blood samples are collected pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 12, 24, 36, 48, 72 and 96 hours post dose
  Samples taken during each of the 6 treatments
Pharmacokinetics of selumetinib by assesement of apparent volume at distribution steady state, (MRT)*CL/F (Vss/F) | Blood samples are collected pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 12, 24, 36, 48, 72 and 96 hours post dose
  Samples taken during each of the 6 treatments
Pharmacokinetics of selumetinib by assesement of apparent volume at distribution (Vz/F) | Blood samples are collected pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 12, 24, 36, 48, 72 and 96 hours post dose
  Samples taken during each of the 6 treatments
Pharmacokinetics of selumetinib and N-desmethyl selumetinib by assesement of terminal half-life (t1/2) | Blood samples are collected pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 12, 24, 36, 48, 72 and 96 hours post dose
  Samples taken during each of the 6 treatments
Pharmacokinetics of selumetinib and N-desmethyl selumetinib by assesement of terminal rate constant (λz) | Blood samples are collected pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 12, 24, 36, 48, 72 and 96 hours post dose
  Samples taken during each of the 6 treatments
Pharmacokinetics of selumetinib and N-desmethyl selumetinib by assesement of AUC metabolite to parent ratio (MRAUC) | Blood samples are collected pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 12, 24, 36, 48, 72 and 96 hours post dose
  Samples taken during each of the 6 treatments
Pharmacokinetics of selumetinib and N-desmethyl selumetinib by assesement of Cmax metabolite to parent ratio (MRCmax) | Blood samples are collected pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 12, 24, 36, 48, 72 and 96 hours post dose
  Samples taken during each of the 6 treatments
Pharmacokinetics of selumetinib by assesement of mean residence time (MRT) | Blood samples are collected pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 12, 24, 36, 48, 72 and 96 hours post dose
  Samples taken during each of the 6 treatments

OTHER OUTCOMES:
Safety variables (adverse events, physical examinations, opthalmologic assessements, vital signs, clinical laboratory assessments and 12 lead electrocardiograms) | Baseline (Day-1) up to Day 24
  Assessments performed during each of the 6 treatments

CONTACTS AND LOCATIONS:
Overall Officials: David R Mathews, MD, Principal Investigator — Quintiles 6700 W 115th Street, Kansas, US
Locations (1):
- Research Site, Overland Park, Kansas, United States

REFERENCES:
- See also: CSR_Synopsis_D1532C00083 — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=2514&filename=CSR_Synopsis_D1532C00083.pdf